CLINICAL TRIAL: NCT02840149
Title: Correlation Between SUV on 68Ga-DOTATATE PET/CT and Ki-67 Index in Neuro-Endocrine Tumors
Brief Title: SUV on 68Ga-DOTATATE PET/CT and Ki-67 Index in Neuro-Endocrine Tumors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Gad Abikhzer, MD, Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CODIM-MDM-16-211
Record Dates: First submitted 2016-07-14; First posted 2016-07-21 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2023-12

CONDITIONS: Neuroendocrine Tumors
Keywords: 68Ga-DOTA-TATE, PET/CT
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga-DOTATATE PET/CT (Other): 68Ga-DOTATATE PET/CT scan performed on Neuro-endocrine tumor patients
  Interventions: Drug: 68Ga-DOTATATE PET/CT

INTERVENTIONS:
Drug: 68Ga-DOTATATE PET/CT — 68Ga-DOTATATE PET/CT scan

SUMMARY:
Positron emission tomography/computed tomography (PET/CT) is an advanced nuclear medicine scan. This technology allows precise and early cancer to be visualized and measured on whole body images. Patients with Neuro-Endocrine tumors (NETs), require specialized molecular imaging to stage, re-stage and assess eligibility and response to therapy. 68Ga-DOTATATE is a nuclear medicine imaging agent that is not yet approved by Health Canada but used extensively throughout the world. The Ki-67 index, a marker of cell proliferation in NETs, is one of the most important prognostic factors in this disease. The objective of this study is to evaluate if the maximal standard uptake value (SUVmax) on PET/CT in NETs inversely correlates with Ki-67 score on initial biopsy. If this hypothesized correlation between SUV and Ki-67 score is reproduced, then DOTATATE would serve as a non-invasive method to assess cellular proliferation and therefore prognosis of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Known or suspected somatostatin receptor positive tumor such as: neuroendocrine tumor (carcinoid, gastro-entero-pancreatic neuroendocrine tumors, etc); pheochromocytoma; neuroblastoma; medulloblastoma; ectopic Cushing syndrome/non-pituitary ACTH elevation; tumor-induced osteomalacia. Supporting evidence may include MRI, CT, biochemical markers, and/or pathology report.
* Previous diagnosis of NET with Ki-67 index available or soon to be obtained.
* ECOG performance status 0 - 3, inclusive.
* 18 years or older and able to understand and provide written informed consent
* Patients must be able to tolerate the physical/logistical requirements of a PET/CT scan including lying supine for up to 45 minutes with the arms above the head and tolerating intravenous cannulation for injection of the study drug

Exclusion Criteria:

* Medically unstable patients (e.g. acute cardiac or respiratory distress or hypotensive, etc.)
* Patients who exceed the safe weight limit or bore of the PET/CT bed
* Patients who are claustrophobic or pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Correlation between SUV on 68Ga-DOTATATE PET/CT with Ki-67 index in NET | 2 years
  To determine whether there is an inverse correlation between SUV on 68Ga-DOTATATE PET/CT with Ki-67 index in patients with neuroendocrine tumors

CONTACTS AND LOCATIONS:
Overall Officials: Gad Abikhzer, MDCM, Principal Investigator — McGill University Health Centre, Jewish General Hospital; Stephan Probst, MDCM, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No